CLINICAL TRIAL: NCT03168022
Title: A SINGLE-DOSE, RANDOMIZED, OPEN-LABEL, TWO-WAY CROSSOVER BIOEQUIVALENCE STUDY OF TNX-102 SL (CYCLOBENZAPRINE HCL SUBLINGUAL TABLETS) 2.8 mg FROM TWO MANUFACTURERS IN HEALTHY SUBJECTS UNDER FASTING CONDITIONS
Brief Title: Bioequivalence Study of TNX-102 SL 2.8 mg Sublingual Tablets From Two Manufacturers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TNX-CY-F105
Record Dates: First submitted 2017-04-25; First posted 2017-05-30 (Actual); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Healthy Adults
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Treatment A (Experimental): 1 x TNX-102 SL 2.8 mg yellow tablet (commercial manufacturer) to be held under the tongue until dissolved.
  Interventions: Drug: Treatment A
- Treatment B (Experimental): 1 x TNX-102 SL 2.8 mg white tablet (original manufacturer) to be held under the tongue until dissolved.
  Interventions: Drug: Treatment B

INTERVENTIONS:
Drug: Treatment A — 1 x TNX-102 SL 2.8 mg yellow tablet (commercial manufacturer) to be held under the tongue until dissolved.
  Other Names: cyclobenzaprine HCl
  Arms: Treatment A
Drug: Treatment B — 1 x TNX-102 SL 2.8 mg white tablet (original manufacturer) to be held under the tongue until dissolved.
  Other Names: cyclobenzaprine HCl
  Arms: Treatment B

SUMMARY:
This study is an open-label, 2-way crossover, single-dose study that is being performed to establish the bioequivalence of TNX-102 SL 2.8 mg tablets from two manufacturers: manufacturer of the Phase 2/3 drug product and manufacturer of the Phase 3 and commercial drug product. This bioequivalence study will confirm (1) the drug product manufactured from these two manufacturers are therapeutically equivalent and (2) the efficacy and safety data obtained in clinical studies using TNX-102 SL from these two manufacturers are comparable.

DETAILED DESCRIPTION:
This will be a single centre, bioequivalence, open-label, randomized, single-dose, 2-period, 2 sequence, crossover study under fasting conditions.

Potential subjects will be screened by medical and psychiatric history, and laboratory and physical examinations 2 to 30 days prior to drug administration. All eligible subjects will be admitted to the study unit on Day -1, the day prior to dose administration. Baseline values will be considered the last value obtained before dosing for each assessment. On Day 1, the morning after admission, after all pre-dose assessments have been completed and subjects who remain eligible have agreed to continue, subjects will be randomly assigned to study medication and will receive the assigned test drug. Subjects will be required to fast for at least 10 hours prior to dosing until at least 4 hours post-dose.

For each period, subjects will be confined to the study site from at least 10 hours before dosing until after the 24-hour post-dose blood draw. Subjects will come back for all subsequent blood draws. Subjects will be reassessed for eligibility prior to each dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between 18 and 65 years of age, non-smoker.
2. Body mass index >18.5 and <30.0 kg/m2
3. Females of childbearing potential must be willing to use a medically acceptable method of birth control throughout the study.
4. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening
2. Positive hepatitis B, hepatitis C, HIV, urine drug screen, urine cotinine test, or alcohol breath test at screening.
3. History of hypersensitivity to cyclobenzaprine, any of the formulation component, or other related drugs.
4. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration.
5. Positive pregnancy test at screening.
6. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities at screening.
7. History of significant alcohol or drug abuse within one year prior to screening
8. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
9. Use of medication other than topical products without significant systemic absorption and hormonal contraceptives
10. Breast-feeding subject.
11. Presence of dentures, tongue piercings with ongoing use of tongue studs/jewelry, orthodontic braces, or surgical manipulations of the tongue.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Audet, MD, Principal Investigator — inVentiv
Locations (1):
- InVentiv Health Clinique Inc., Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A First, Then B: Single Dose of Treatment A (TNX-102 SL 2.8 mg yellow tablet [commercial manufacturer]), Washout 21 days, Single Dose of Treatment B (TNX-102 SL 2.8 mg white tablet [original manufacturer])
- Treatment B First, Then A: Single Dose of Treatment B (TNX-102 SL 2.8 mg white tablet [original manufacturer]), Washout 21 days, Single Dose of Treatment A (TNX-102 SL 2.8 mg yellow tablet [commercial manufacturer])
Period: Overall Study
Arm/Group | Treatment A First, Then B | Treatment B First, Then A
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All subjects that were randomized to receive all treatments.
Arm/Group | All Study Participants
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Concentration (AUC) of Cyclobenzaprine
Description: Blood samples were collected prior to drug administration and 0.083 (5 min), 0.167 (10 min),0.333 (20 min), 0.500 (30 min), 0.750 (45 min), 1.00, 1.50, 2.00, 2.50, 3.00, 3.33, 3.67, 4.00, 4.33, 4.67, 5.00, 5.50, 6.00, 8.00, 12.0, 16.0, 24.0, 36.0, 48.0, 72.0, and 96.0 hours post-dose in each period.
Time Frame: 0 to 96 hours
Population: Subjects who completed the study and for whom the PK profile could be adequately characterized were included in the outcome measures.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Groups:
- Treatment A: All study subjects who were administered one TNX-102 SL 2.8 mg yellow tablet (commercial manufacturer) under fasting conditions and completed the study.
- Treatment B: All study subject who were administered one TNX-102 SL 2.8 mg white tablet (original manufacturer) under fasting conditions and completed the study.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
pg*h/mL | 70066.90 (25158.61) | 64711.53 (22633.07)

2. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) of Treatment A and Treatment B, Administered as 1 x 2.8 mg TNX-102 SL Under Fasting Conditions.
Description: The MedDRA® dictionary was used to classify all TEAEs reported during the study by System Organ Class (SOC) and Preferred Term (PT).
Time Frame: Continuously until the end (day 5) of each study period + 8-10 days after end of last period (total duration: about 1 month)
Population: All subjects who received at least one dose of either Treatment A or Treatment comprised the safety population (N = 43). Of these, 1 subject discontinued from the study after one dose of Treatment B and was replaced with a stand-by. A total 42 subjects completed the study as per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 43
Participants | 18 | 19

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 13.
Groups:
- Treatment A: All subjects who were administered TNX-102 SL 2.8 mg yellow tablet (commercial manufacturer).
- Treatment B: All subjects who were administered TNX-102 SL 2.8 mg white yellow tablet (original manufacturer).
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 18/42 | 19/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=42) | Treatment B (N=43)
Hypoaesthesia oral (Gastrointestinal disorders) | 13 | 13
Somnolence (Nervous system disorders) | 5 | 4
Product taste abnormal (General disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days